CLINICAL TRIAL: NCT06325722
Title: Diet Order Effects of Low Fat vs. Low Carb Diets on Body Fat Change
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 10001680; 001680-DK
Record Dates: First submitted 2024-03-21; First posted 2024-03-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-15

CONDITIONS: Overweight; Obesity
Keywords: Diet; Body Fat; Nutrition; weight-loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-carbohydrate diet then low-fat diet (Experimental): A low-carbohydrate followed by low-fat diet, each lasting for 4 weeks in adults with overweight or obesity
  Interventions: Other: Low-carbohydrate Diet; Other: Low-fat Diet
- low-fat diet then low-carbohydrate diet (Experimental): A low-fat followed by low-carbohydrate diet, each lasting for 4 weeks in adults with overweight or obesity
  Interventions: Other: Low-carbohydrate Diet; Other: Low-fat Diet

INTERVENTIONS:
Other: Low-carbohydrate Diet — Consisting of 15 percent protein, 75 percent fat, and 10 percent carbohydrate
Other: Low-fat Diet — Consisting of 15 percent protein, 10 percent fat, and 75 percent carbohydrate

SUMMARY:
Background:

In a previous study, participants were lived at the NIH and randomly received either a low-fat or a low-carbohydrate diet for 2 weeks and then switched to the other diet for 2 more weeks. Participants who received the low-carbohydrate diet first lost more body fat at the end of the study than those who received the low-fat diet first. Researchers want to see if they can repeat that result in a longer weight loss study when participants live at home.

Objective:

To test the effects of diet order in people receiving either a low-fat or low-carbohydrate diet first for 4 weeks and then immediately switched to the other diet for another 4 weeks.

Eligibility:

Adults aged 19 to 50 years with a body mass index of 25 or more.

Design:

Participants will complete the study at their homes, but there will be 3 required visits to the NIH. Participants will drink a special type of water 2 weeks before the baseline NIH visit and collect urine samples at home to measure how many calories they burn. Before the diets begin, participants will visit the NIH for baseline testing when they will have a metabolism test while relaxing in a bed with a plastic hood over their head to collect the air they breathe out. They will have scans to measure their bone density and how much muscle and body fat they have. They will give stool, blood, and urine samples.

Participants will be asked to eat a specific diet for 4 weeks followed by a different diet for 4 weeks. All meals will be delivered to the participants' homes. They will eat only the foods delivered.

Participants will weigh themselves daily. They will wear a monitor to track their physical activity and a sensor to measure their glucose levels. They will prick their finger each morning to test a drop of blood for ketones. Participants will meet virtually as a group with the study team weekly. Participants will have two more NIH visits towards the end of each diet period....

DETAILED DESCRIPTION:
Study Description:

This is an 8-week crossover outpatient feeding trial of a low carbohydrate versus a low-fat diet, each provided for 4 weeks in random order with no washout period, in adult volunteers with overweight or obesity.

Objectives:

Primary Objectives: To determine the effect of diet order on the mean total fat mass change in subjects randomized to receive either a low carbohydrate followed by a low fat diet or the reverse order, with each diet lasting for 4 weeks.

Secondary Objectives: To determine the effect of diet order on the mean rate of body weight change in subjects randomized to receive either a low carbohydrate followed by a low fat diet or the reverse order, with each diet lasting for 4 weeks and the rate of weight change is measured during the last 2 weeks of each diet. To determine the effect of diet order on mean total body weight change in subjects randomized to receive either a low carbohydrate followed by a low fat diet or the reverse order, with each diet lasting for 4 weeks.

Endpoints:

Primary Endpoint: Mean total fat mass change measured by dual energy X-ray absorptiometry at baseline and week 8.

Secondary Endpoints: Mean rate of weight change by linear mixed modeling of daily weight measurements. Mean total body weight change measured between baseline and week 8.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Adults aged 18-50 years
3. Weight stable (< +/- 5 percent over past 6 months) as determined by volunteer report
4. Body mass index (BMI) >= 25 kg/m^2
5. Agreement to adhere to Lifestyle Considerations throughout the study duration

EXCLUSION CRITERIA:

1. Subjects with cardiac pacemakers or other implants that may be affected by or affect the DXA measurements
2. Inadequate access to equipment required for the study (e.g., too little refrigerator storage space or a microwave oven that is too small) as determined by discretion of PI and/or study team
3. Evidence of diseases or conditions that may influence appetite (e.g., cancer, diabetes, alterations of smell or taste post COVID-19), diseases or conditions that affect the immune system, or other conditions at the discretion of the PI and/or study team
4. Taking prescription medications or other drugs that may influence metabolism (including but not limited to diet/weight-loss medication, some psychiatric medications, or other medications at the discretion of the PI and/or study team)
5. People unlikely to adhere to a relatively consistent daily and weekly routine and avoid travel during their participation in the study. For example, people with occupations such as pilots, flight attendants, or frequently travel for work or pleasure.
6. People unlikely to abstain from off study food or supplements that may impact metabolism or appetite at the discretion of the study team
7. Positive pregnancy test or lactating as determined by volunteer report (women only)
8. Inability or unwillingness to use birth control between screening and completion of the study (women only)
9. Symptoms or signs of perimenopause or menopause by volunteer report (women only)
10. Regular vigorous exercise >150 min per week as determined by volunteer report
11. Alcohol consumption > 3 drinks per day as determined by volunteer report
12. Regular use of tobacco (smoking, chewing, or vaping), nicotine replacement therapy, or illicit drugs over past 6 months as determined by volunteer report. Subjects may also be excluded based on a urine drug test.
13. Psychological conditions as determined by DSM-5 Self-rated Level 1 Cross-cutting Symptom Measure such as (but not limited to) eating disorders, depression, bipolar disorders, that would be incompatible with safe and successful participation in this study, as determined by investigators
14. Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, food allergies) or a reported dislike of a significant fraction of the study foods
15. Volunteers unwilling or unable to give informed consent
16. Non-English speakers due to unavailability of required questionnaires in other languages

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in total fat mass | 8 weeks
  Change in total fat mass (kg) as measured by dual energy X-ray absorptiometry (DXA) from baseline to week 8

SECONDARY OUTCOMES:
Rate of body weight change from baseline to week 8 | 8 weeks
  Rate of body weight change (kg/d) from baseline to week 8
Rate of body weight change during low-carbohydrate diet | Last 2 weeks of low-carbohydrate diet period
  Rate of body weight change (kg/d) during the last two weeks of the low-carbohydrate diet
Rate of body weight change during low-fat diet | Last 2 weeks of low-fat diet period
  Rate of body weight change (kg/d) during the last two weeks of the low-fat diet

CONTACTS AND LOCATIONS:
Overall Officials: Valerie L Darcey, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Body fat and body weight data
Supporting Information: Study Protocol, Analytic Code
Time Frame: Upon publication in peer reviewed journal
Access Criteria: Open, general access

REFERENCES:
- [Background] Sciarrillo CM, Guo J, Hengist A, Darcey VL, Hall KD. Diet order affects energy balance in randomized crossover feeding studies that vary in macronutrients but not ultra-processing. medRxiv [Preprint]. 2023 Oct 4:2023.10.03.23296501. doi: 10.1101/2023.10.03.23296501. PMID 37986904
- [Background] Hall KD, Guo J, Courville AB, Boring J, Brychta R, Chen KY, Darcey V, Forde CG, Gharib AM, Gallagher I, Howard R, Joseph PV, Milley L, Ouwerkerk R, Raisinger K, Rozga I, Schick A, Stagliano M, Torres S, Walter M, Walter P, Yang S, Chung ST. Effect of a plant-based, low-fat diet versus an animal-based, ketogenic diet on ad libitum energy intake. Nat Med. 2021 Feb;27(2):344-353. doi: 10.1038/s41591-020-01209-1. Epub 2021 Jan 21. PMID 33479499
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001680-DK.html